CLINICAL TRIAL: NCT03323970
Title: Decision Making in Neonatology : a Qualitative Study
Acronym: PRODA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2014/219
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians
  Interventions: Other: semi-structured interviews

INTERVENTIONS:
Other: semi-structured interviews — individual semi-structured interviews

SUMMARY:
This study aimed to describe and understand the decision making process in neonatology in situations of limiting of withdraw life sustaining treatments, by conducting interviews with physicians from one neonatology unit.

ELIGIBILITY:
Inclusion Criteria:

* Physicians in charge of new born babies for whom a decision making regarding limiting or withdrawing treatments is emerging.
* physicians' informed consent to participate to an interview
* parents' informed consent to collect data concerning their new born.

Exclusion Criteria:

- Not fluent French speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study concerns the situation of new born for whom a decision making regarding limiting or withdrawing treatments is emerging, but only the physicians are involved as subjects of the study and seen in interviews.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
semi-structured interviews | 3 months
  qualitative data analysis - theorical saturation

IPD SHARING:
Plan to Share IPD: No